CLINICAL TRIAL: NCT07201519
Title: Phase IIa Study of Safety/Feasibility of a Hybrid Model of Tertiary and Community Delivery of Hepatic Artery Infusion Chemotherapy
Brief Title: Study of Safety/Feasibility of a Hybrid Model of Tertiary and Community Delivery of Hepatic Artery Infusion Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael J Cavnar, MD (Other)
Responsible Party: Sponsor-Investigator, Michael J Cavnar, MD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102585
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer Metastatic; Intrahepatic Cholangiocarcinoma
Keywords: hepatic artery infusion; chemotherapy; floxuridine
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Community Mental Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tertiary Oncology Cohort (TO) (Active Comparator): receive care as per usual institutional protocol, visits every two weeks and standard manual HAI dose calculation.
  Interventions: Device: Hepatic Artery Infusion Pump (HAIP); Procedure: Standard Treatment; Drug: Systemic Chemotherapy Standard of Care; Drug: Standard Of Care targeting driver mutations
- Community Oncology Cohort (CO) (Experimental): HAI pump fills in home by a home infusion company; systemic therapy treatments at the community oncology office; oversight via telehealth visits
  Interventions: Device: Hepatic Artery Infusion Pump (HAIP); Procedure: Community Treatment; Drug: Systemic Chemotherapy Standard of Care; Drug: Standard Of Care targeting driver mutations

INTERVENTIONS:
Device: Hepatic Artery Infusion Pump (HAIP) — HAIP will be filled with mixture of FUDR + Dexamethasone, Heparin & Saline for a 14 day infusion of drugs, followed by a 14 day infusion of Heparin+Saline.
  Other Names: Intera 3000
Procedure: Standard Treatment — systemic therapy per standard-of-care and institutional standards; visits every two weeks and standard manual HAI dose calculation
  Other Names: Tertiary Oncology (TO)
  Arms: Tertiary Oncology Cohort (TO)
Procedure: Community Treatment — systemic therapy fill by home infusion based on TO orders. In person visit with CO for systemic chemotherapy with dose recommendations from TO. Locally obtained testing with telehealth visits with TO team.
  Other Names: Community Oncology (CO)
  Arms: Community Oncology Cohort (CO)
Drug: Systemic Chemotherapy Standard of Care — Dosing of systemic therapy will be according to established routine practice guidelines. Patients with colon cancer will receive systemic chemotherapy that will consist of either FOLFIRI, FOLFOX, or Irinotecan/oxaliplatin at the discretion of the oncologist.
  Patients with intrahepatic cholangiocarcinoma will receive Gemcitabine/Oxaliplatin or Gemcitabine alone, at the discretion of the oncologist.
Drug: Standard Of Care targeting driver mutations — Per current SOC guidelines, EGFR inhibitors targeting driver mutations (e.g., RAS wild-type) will be administered as appropriate (FDA-approved agents such as Panitumumab for EGFR)

SUMMARY:
The goal of this clinical trial is to help learn about the safety and feasibility of hepatic artery infusion chemotherapy for those who have colorectal liver metastases, both resectable and unresectable, or unresectable intrahepatic cholangiocarcinoma. The main questions it aims to answer are:

* safety and feasibility of installing a pump that deliveries chemotherapy to the hepatic artery (the blood vessel that supplies blood to the liver)
* help learn more about the safety of patients having pump refills at home or a local clinic versus having it routinely done at the hospital

Participants will have surgery to install a pump which is a standard surgical procedure. After surgery, participants will select to either receive treatment at the hospital facility or with a community oncologist that will provide cancer care to participants close to home, rather than in a large hospital or academic medical center.

The main treatment on study will last about 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal adenocarcinoma metastatic to the liver which is either Unresectable (group A) or Resectable (group B; ie, will be completely resected), AND with no definitive clinical or radiographic evidence of extrahepatic disease other than: metastatic disease to resectable peri-hepatic lymph nodes; up to 5 proven or suspected lung metastases, provided they are stable or responding in number and size for a minimum of 2-months of systemic chemotherapy and are amenable to SBRT or resection. or
* Histologically confirmed unresectable intrahepatic cholangiocarcinoma (group C), with presence of less than 70% liver involvement with no definitive clinical or radiographic evidence of extrahepatic metastatic disease other than resectable perihepatic lymph nodes.
* Patients > or equal 18 years of age
* ECOG Performance Status of 0 - 1 (APPENDIX C)
* Lab Values < or equal 14 days prior to study enrollment: absolute neutrophil count > or equal 1,500/mcL Total Bilirubin < or equal 1.5 mg/dL AST/ALT < 5 x institutional upper limit of normal (ULN) Platelets > or equal 100,000/mcL Creatinine < 1.5 mg/dL HGB > 8 g/dL INR < or equal 1.5
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Prior chemotherapy is acceptable if last dose given > or equal 3 weeks prior to study enrollment
* Any investigational agent is acceptable if last dose administered > or equal 3 months before study enrollment
* In order for patients to select treatment in the CO arm, they must have the ability to do telehealth visits, either via a home computer, tablet, or smartphone, either via home internet access or cellphone network.

Exclusion Criteria:

* Presence of distant non-liver metastatic disease confirmed by radiographic evaluation. Clinical or radiographic evidence of metastatic disease to regional peri-hepatic lymph nodes will be allowed, provided it is amenable to resection. For the colorectal carcinoma only: Up to 5 lung metastases are allowable, provided they are stable (or responding) in number and size for minimum of 2-mos of systemic chemo and are amenable to SBRT.
* Microsatellite instability (MSI) or Mismatch repair deficiency (MMR-D)
* Prior radiation to the liver, including external beam, SBRT, Y90. Prior radiation therapy to the pelvis is acceptable
* Bevacizumab (Avastin®) cannot be given concurrently with HAI FUDR. Patients can previously have received it with a minimum 6-week washout period
* Active infection, hepatic encephalopathy
* Clinical evidence of portal hypertension (ascites, gastroesophageal varices or portal vein thrombosis) are exclusions. Note: surgically-related ascites does not exclude the patient.
* Female patients who are pregnant or lactating - or planning to become pregnant within 6 months after the end of the treatment (female patients of childbearing potential must have negative pregnancy test prior to surgery)
* If in the opinion of the treating investigator a patient has any serious medical problems which may preclude receiving this type of treatment
* Patients with history or known presence of primary CNS tumors, seizures not well-controlled with standard medical therapy; Patients with a history of stroke within 3 months or with substantial residual deficit, based on investigator discretion
* Serious or non-healing active wound, ulcer, or bone fracture
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the HAIP chemotherapy (i.e., investigational regimen)
* Patients with psychiatric illness or social situations that would limit compliance with study requirements. Examples: active substance abuse, active severe alcohol abuse, etc.
* Inability to reliably commit to traveling to either Lexington, KY (for patients choosing TO site for HAI administration) or local CO site every 2 weeks for duration of the study treatment (6 months). Patient must have readily identifiable, reliable primary and back-up modes of transportation regardless of weather.
* Patients with AXIOS™ stents (or similar) used to connect the small intestine to the gastric remnant after a prior gastric bypass for access for ERCP/stent in the setting of biliary obstruction are eligible at the discretion of the investigator. Considerations regarding eligibility comprise removal of the stent prior to HAIP implantation, or the placement of the HAIP catheter at least 5cm away from the AXIOS stent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with HAI Pump still in use at 3 months | 3 months
  The primary outcome is safety, defined as: continued functional / in-use HAI pump (either for FUDR fills or maintenance saline/glycerine fills) at 3-months.

SECONDARY OUTCOMES:
Number of Adverse events according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 4 months
Number of participants transferring care | 3 months
  Determine the number of Community Oncology (CO) HAI patients that permanently transfer their care to tertiary center due to CO access issues or other reasons
Number of administered HAI cycles | 1 year
  Tabulate the number of administered HAI cycles at 1-year post-enrollment
Number of failed access visits by home infusion | 3 months
  Home infusion HAI access issues for Cycles 1 - 3, assessed by the number of failed access visits by home infusion requiring a trip to the institution for pump access/troubleshooting
Number of participants with biliary sclerosis | 1 year
  biliary sclerosis is determined by the treating physician
Number of participants with biliary sclerosis | 2 years
  biliary sclerosis is determined by the treating physician
Overall Response Rate (via RECIST v1.1) | 3 months
  In patients with measurable disease (unresectable CLM and unresectable intrahepatic cholangiocarcinoma, measure Overall Response Rate (via RECIST v1.1) to standard hepatic artery infusion chemotherapy (FUDR) combined with standard systemic chemotherapy (tailored to primary disease), and conversion to resection at 1-year post-study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cavnar, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No